CLINICAL TRIAL: NCT05470764
Title: Randomized, Open-label, Single-dose, Two-sequence, Two-period, Crossover, Comparative, Oral Bioequivalence Study of Test Product PERINDOPRES® TRIO, 8 mg Perindopril Tert-Butylamine / 2.5 mg Indapamide/ 10 mg Amlodipine Tablets (PrJSC "Pharmaceutical Firm "Darnitsa") And Reference Product TRIPLIXAM® 10 mg /2.5 mg/10 mg, 10 mg Perindopril Arginine / 2.5 mg Indapamide / 10 mg Amlodipine Film-Coated Tablets (Manufactured By Servier (Ireland) Industries Ltd) In Healthy, Adult Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of 8 mg Perindopril Tert-Butylamine / 2.5 mg Indapamide / 10 mg Amlodipine Tablets Versus 10 mg Perindopril Arginine / 2.5 mg Indapamide / 10 mg Amlodipine Film-Coated Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Darnitsa Pharmaceutical Company (Industry)
Collaborators: International Pharmaceutical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PER02-E
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Bioequivalence; Healthy Subjects
Keywords: bioequivalence; perindopril; indapamide; amlodipine; healthy subjects; pharmacokinetics
MeSH Terms: interventions — perindopril tert-butylamine; Indapamide; Amlodipine

STUDY DESIGN:
Intervention Model Description: Two-period, two-sequence, cross-over single dose study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PERINDOPRES® TRIO (Test) (Experimental): A single oral dose of the test product PERINDOPRES® TRIO 8 mg perindopril tert-butylamine / 2.5 mg indapamide / 10 mg amlodipine tablets.
  Interventions: Drug: PERINDOPRES® TRIO, 8 mg perindopril tert-butylamine / 2.5 mg indapamide / 10 mg amlodipine tablets
- TRIPLIXAM® 10 mg /2.5 mg/10 mg (Active Comparator): A single oral dose of the reference product TRIPLIXAM® 10 mg /2.5 mg/10 mg, 10 mg perindopril arginine / 2.5 mg indapamide / 10 mg amlodipine film-coated tablets.
  Interventions: Drug: TRIPLIXAM® 10 mg /2.5 mg/10 mg, 10 mg perindopril arginine / 2.5 mg indapamide / 10 mg amlodipine film-coated tablets

INTERVENTIONS:
Drug: PERINDOPRES® TRIO, 8 mg perindopril tert-butylamine / 2.5 mg indapamide / 10 mg amlodipine tablets — Oral, generic fixed-dose combination of perindopril tert-butylamine (angiotensin-converting-enzyme inhibitor for the treatment of high blood pressure and heart failure), indapamide (thiazide-like diuretic used in the treatment of hypertension and decompensated heart failure) and amlodipine (calcium channel blocker used to treat high blood pressure and coronary artery disease).
  Arms: PERINDOPRES® TRIO (Test)
Drug: TRIPLIXAM® 10 mg /2.5 mg/10 mg, 10 mg perindopril arginine / 2.5 mg indapamide / 10 mg amlodipine film-coated tablets — Oral, innovative fixed-dose combination of perindopril arginine (angiotensin-converting-enzyme inhibitor for the treatment of high blood pressure and heart failure), indapamide (thiazide-like diuretic used in the treatment of hypertension and decompensated heart failure) and amlodipine (calcium channel blocker used to treat high blood pressure and coronary artery disease).
  Arms: TRIPLIXAM® 10 mg /2.5 mg/10 mg

SUMMARY:
The present study is a comparative bioavailability study performed to assess bioequivalence between a Test medication (PERINDOPRES® TRIO, 8 mg perindopril tert-butylamine / 2.5 mg indapamide / 10 mg amlodipine tablets manufactured by PrJSC "Pharmaceutical firm "Darnitsa" [Ukraine]) and a Reference medication (marketed medicinal product TRIPLIXAM® 10 mg /2.5 mg/10 mg, 10 mg perindopril arginine / 2.5 mg indapamide / 10 mg amlodipine film-coated tablets [manufactured by Servier (Ireland) Industries Ltd]) in healthy adult volunteers under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects, age 18 to 50 years, inclusive, body mass index (BMI) range is within 18.5 - 30.0 kg/m2, subject does not have a known allergy to the drug under investigation or any of its ingredients or any other related drugs, standard ECG assessment is normal (no QTc prolongation), medical history and physical examination within medically acceptable criteria, laboratory investigations tests within laboratory reference ranges (ALP and creatinine are accepted if below the reference range after being evaluated by the physician as clinically not significant). Haematology tests within 5% of reference limits.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of perindopril | Blood sampling for pharmacokinetic analysis covered up to 36 hours post-dose
  The Cmax value is based on perindopril plasma concentration.
Area under the concentration-time curve from time zero to the last quantifiable concentration (AUC0-t) of perindopril | Blood sampling for pharmacokinetic analysis covered up to 36 hours post-dose
  The AUC0-t is the area under the plasma concentration versus time curve from time zero (predose) to time of last quantifiable concentration (t) and is based on perindopril plasma concentration.
Cmax of indapamide | Blood sampling for pharmacokinetic analysis covered up to 72 hours post-dose
  The Cmax value is based on indapamide plasma concentration.
AUC0-t of indapamide | Blood sampling for pharmacokinetic analysis covered up to 72 hours post-dose
  The AUC0-t is the area under the plasma concentration versus time curve from time zero (predose) to time of last quantifiable concentration (t) and is based on indapamide plasma concentration.
Cmax of amlodipine | Blood sampling for pharmacokinetic analysis covered up to 72 hours post-dose
  The Cmax value is based on amlodipine plasma concentration.
Area under the concentration-time curve from time zero to 72 hours (AUC0-72) of amlodipine | Blood sampling for pharmacokinetic analysis covered up to 72 hours post-dose
  The AUC0-72 is the area under the plasma concentration versus time curve from time zero (predose) to 72 hours and is based on amlodipine plasma concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- International Pharmaceutical Research Center, Amman, Jordan